CLINICAL TRIAL: NCT05445336
Title: The iCARE Study: An Integrated Collection of Education Modules on Fall and Fracture Prevention for Healthcare Providers
Brief Title: The iCARE Study: Education Modules for Fracture Prevention
Acronym: iCARE
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Alexandra Papaioannou, Executive Director and Clinician Scientist, GERAS Centre for Aging Research, Hamilton Health Sciences Corporation
Other Study IDs: 14463
Record Dates: First submitted 2022-01-28; First posted 2022-07-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2023-12

CONDITIONS: Osteoporosis; Frailty; Chronic Conditions, Multiple; Fracture
Keywords: Frailty; Service Provision; Education; Knowledge Translation; Knowledge Mobilization; Osteoporosis; Fracture Prevention; Long Term Care
MeSH Terms: conditions — Osteoporosis; Frailty; Multiple Chronic Conditions; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Internal Champion & LTC Leadership Team #1 from Site #1: The internal champion and LTC leadership team of each LTC home will attend two virtual focus group sessions to help co-design the PREVENT Program educational material. The internal champion will receive training on how to deliver the PREVENT program to the leadership team. The internal champion/pharmacist/data analyst will receive training on how to develop an audit and feedback report on fall and fracture management. All participants will attend an educational meeting facilitated by the internal champion who will use a combination of didactic and interactive activities. After the educational meeting, the leadership team will complete an action and care planning report for each LTC resident at high risk of fracture. Lastly, all participants will attend two virtual focus group sessions to discuss the successes and challenges of implementing the PREVENT program in practice.
  Interventions: Behavioral: PREVENT Program
- Internal Champion & LTC Leadership Team #2 from Site #2: The internal champion and LTC leadership team of each LTC home will attend two virtual focus group sessions to help co-design the PREVENT Program educational material. The internal champion will receive training on how to deliver the PREVENT program to the leadership team. The internal champion/pharmacist/data analyst will receive training on how to develop an audit and feedback report on fall and fracture management. All participants will attend an educational meeting facilitated by the internal champion who will use a combination of didactic and interactive activities. After the educational meeting, the leadership team will complete an action and care planning report for each LTC resident at high risk of fracture. Lastly, all participants will attend two virtual focus group sessions to discuss the successes and challenges of implementing the PREVENT program in practice.
  Interventions: Behavioral: PREVENT Program
- Internal Champion & LTC Leadership Team #3 from Site #3: The internal champion and LTC leadership team of each LTC home will attend two virtual focus group sessions to help co-design the PREVENT Program educational material. The internal champion will receive training on how to deliver the PREVENT program to the leadership team. The internal champion/pharmacist/data analyst will receive training on how to develop an audit and feedback report on fall and fracture management. All participants will attend an educational meeting facilitated by the internal champion who will use a combination of didactic and interactive activities. After the educational meeting, the leadership team will complete an action and care planning report for each LTC resident at high risk of fracture. Lastly, all participants will attend two virtual focus group sessions to discuss the successes and challenges of implementing the PREVENT program in practice.
  Interventions: Behavioral: PREVENT Program

INTERVENTIONS:
Behavioral: PREVENT Program — PREVENT (Person-centred Routine Fracture PreEVENTion) is a scalable model for delivering routine assessments and interventions on diet and supplements, multifactorial fall and fracture prevention strategies, and medications to long term care teams to treat residents at high risk of fracture.

SUMMARY:
A large proportion of older adults living in long term care homes are frail and have osteoporosis. With age, there is a gradual and progressive decline in bone quality and quantity and an increase in frailty, which is associated with increased fracture risk. Additionally, fractures pose a significant burden to the health and quality of life of long term care residents and contribute to high healthcare costs. Despite the high prevalence of osteoporosis, falls, and fractures in long term care, the management of osteoporosis is not optimal among long term care residents at risk of fracture. The aim of this study is to co-design a service provision (i.e., PREVENT - Person-centred Routine Fracture PreEVENTion) with healthcare providers in long term care and to determine the feasibility of implementing PREVENT in long term care settings.

DETAILED DESCRIPTION:
Fractures pose a significant burden on health, quality of life, and mortality of older adults in long term care (LTC) and contribute to high health care costs. PREVENT (Person-centred Routine Fracture PreEVENTion) is a scalable model for delivering routine assessments and interventions on diet and supplements, multifactorial fall and fracture prevention strategies, and medications to long term care teams to treat residents at high risk of fracture. The purpose of the iCARE study is to create a fall and fracture educational program (i.e., PREVENT) for LTC healthcare providers to deliver routine assessments for the management and treatment of osteoporosis. The benefit of such a guide may help to reduce the devastating impact of fractures in older adults residing in LTC homes. The aim of this pilot study is to: 1) determine feasibility and 2) adaptations through facilitators and barriers. Before a larger trial can be implemented to determine the effectiveness of the PREVENT Program in practice, the iCARE study seeks to determine the feasibility of implementing PREVENT in practice and identify strategies to tailor the program to the individual long term care home and care team through design thinking solutions.

ELIGIBILITY:
Organizational Level Inclusion Criteria:

Five long LTC homes in Ontario that

* Have a minimum of 70 residents
* Are publicly owned and private for-profit and private not-for-profit homes in both urban and rural sites

Individual Level Inclusion Criteria:

* At least one internal champion
* Five Professional Advisory Committee (PAC) care teams from five long term care homes in Ontario that provide osteoporosis care to residents.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Care planning in long term care is a collaborative effort between the resident, the long term care healthcare provider, and the resident's family/caregiver. An internal champion will be identified to represent several long term care homes and who will help identify the five Professional Advisory Committees care teams who are the end-users of the PREVENT program. The Professional Advisory Committee may consist of a Director of Care/Nursing Director, Medical Director, Clinical Consultant Pharmacist, and other participating members who may include dietitians, rehabilitation staff, nurses, physicians, and personal support workers.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment Rate | 2 months
  Number of long term care homes (LTCs) in Ontario recruited within two months. Criteria for success: recruit 5 LTC homes in Ontario within 2 months
Feasibility - LTC home readiness and capacity | 1 month
  Determine long term care home readiness and capacity to participate in the iCARE study based on a Readiness Checklist Survey. Criteria for success: at least 75% of homes approached are ready and have the capacity to participate in the study
Feasibility - Length of time to complete PREVENT Program | 4 months
  Length of time for participants to implement the PREVENT Program
Feasibility - Logistics of linking data (Yes/No format) | 4 months
  Determine the logistics of linking MDS 2.0 data with pharmaceutical database data at the resident level. This will be assessed by a "yes" or "no" (i.e., Feasible - Yes vs. Feasible - No)
Fidelity of delivering the PREVENT program | 4-6 months
  Determine the fidelity of delivering the PREVENT program. Criteria for success: ≥ 80% on the fidelity checklist.
Feasibility - Number of Questions Completed | 4 months
  The number of questions answered by the participants for each questionnaire. Criteria for success is 80% of questions are completed.

SECONDARY OUTCOMES:
Changes in Prescribing Habits | 4-6 months
  To determine if appropriate prescribing habits change after the educational session. The criteria for success is a 10% improvement in prescribing habits. This will be measured by the number of prescriptions per number of residents at high risk of fracture pre- vs. post-intervention.
Adaptations to PREVENT Program | 4-6 months
  To determine adaptations to the PREVENT program by facilitating two 1.5-hour focus group sessions (semi-structured interviews) with the leadership team to 1) discuss facilitators of and barriers to implementing the PREVENT program and 2) make necessary changes to the PREVENT program/educational material catered to the individual LTC home.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, MD, MSc, FRCP(c), FACP, Principal Investigator — McMaster University
Locations (1):
- GERAS Centre for Aging Research, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No